CLINICAL TRIAL: NCT05662228
Title: Mechanistic Investigation of Therapies for Down Syndrome Regression Disorder
Brief Title: Therapies for Down Syndrome Regression Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1992
Record Dates: First submitted 2022-12-08; First posted 2022-12-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome; Regression
Keywords: Catatonia; Autoimmune disorder; Sleep; Loss of skills; Autoimmune Encephalopathy
MeSH Terms: conditions — Down Syndrome; Catatonia; Autoimmune Diseases; Autoimmune Diseases of the Nervous System | interventions — Lorazepam; Immunoglobulins, Intravenous; tofacitinib

STUDY DESIGN:
Intervention Model Description: We will use covariate-adaptive randomization to assign participants to one of three treatment arms while accounting for sex, age, and other medical history.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lorazepam (Experimental): Participants will receive lorazepam as an oral pill three times daily for 12 weeks as well as titration doses for an additional 4 weeks (approximately).
  Interventions: Drug: Lorazepam
- Intravenous immunoglobulin (IVIG) (Experimental): Participants will receive 4 doses of IVIG treatment over 12 weeks.
  Interventions: Drug: Intravenous immunoglobulin (IVIG)
- Tofacitinib (Experimental): Tofacitinib will be administered as an oral pill at 5 mg twice daily over the 12-week study.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Lorazepam — Lorazepam will be administered as an oral pill over the first 15 days of study in a daily titration, starting at 0.5 mg BID and increasing to up to 2 mg three times daily, as tolerated. Dosing will continue at the maximum tolerated dose through the 12-week endpoint. Participants will be titrated off lorazepam over at least four weeks after completing the endpoint visit. Taper will be tailored to individuals for safety reasons with a goal of decreasing dosage by 25% weekly. Phone check ins will be conducted every three days to monitor patient.
  Other Names: Ativan
  Arms: Lorazepam
Drug: Intravenous immunoglobulin (IVIG) — IVIG will be administered as a series of four intravenous infusions at a dose of 1 mg/kg with pre-infusion medications of 1 mg/kg diphenhydramine and 15 mg/kg acetaminophen. The first two infusions occur at baseline and one day after (induction dosing), followed by one infusion at 4 weeks and one infusion at 8 weeks.
  Other Names: Gammagard Liquid (immune globulin infusion [human] 10%)
  Arms: Intravenous immunoglobulin (IVIG)
Drug: Tofacitinib — Tofacitinib will be administered as an oral pill at 5 mg twice daily over the 12-week study.
  Other Names: Xeljanz
  Arms: Tofacitinib

SUMMARY:
Individuals with Down syndrome (DS) have an increased risk of numerous co-occurring conditions, including the neuropsychiatric condition known as Down Syndrome Regression Disorder (DSRD). A DSRD diagnosis often includes a sub-acute onset of catatonia, mutism, depersonalization, loss of ability to perform activities of daily living, hallucinations, delusions, and aggression and is most commonly observed in adolescents and young adults.

The study evaluates the safety and efficacy of three currently prescribed therapies: lorazepam, intravenous immunoglobulin (IVIG) and tofacitinib.

DETAILED DESCRIPTION:
Recent published case reports and clinical experience of the investigators indicate Down Syndrome Regression Disorder (DSRD) may be successfully treated with immune-modulating therapies, in addition to current pharmacologic options. This study is a multidimensional clinical trial designed to advance the understanding of the etiology of DSRD and to evaluate the safety and efficacy of three distinct therapeutic approaches to treating DSRD: (1) the benzodiazepine lorazepam (Ativan™) (2) intravenous immunoglobulin (IVIG, Gammagard™) or (3) the JAK inhibitor tofacitinib (Xeljanz™). Participants will be randomized into one of the three treatment arms above for the 12-week study period, with a subset of participants undergoing an initial 12-week observational period.

Specific Aims:

1. To define the relative safety profile of lorazepam, IVIG, and tofacitinib in DSRD.
2. To compare the efficacy of lorazepam, IVIG, and tofacitinib in DSRD.
3. To investigate potential mechanisms underlying DSRD and its response to therapies.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with DS between the ages of 8 and 30 years, inclusive. DS is broadly defined to include complete trisomy 21, Robertsonian translocation trisomy 21, partial trisomy 21 (segmental duplication), and mosaic trisomy 21.
* Diagnosis of possible or probable DSRD per 2022 consensus guidelines.
* Must agree to random treatment assignment.
* Must agree to complete a washout of any medications intended to treat symptoms of DSRD or that may interfere with study interventions.
* Must be able to present with a study partner or legal guardian at all study visits.

Exclusion Criteria:

General

* Weight less than 40 kg.
* Pregnant or breast feeding.
* Past or current tobacco smoking.
* Poor venous access not allowing repeated blood tests or non-compliance with venipuncture requirements.
* Known allergies, hypersensitivity, or intolerance to lorazepam, IVIG, or tofacitinib.
* Participants may be excluded for other unforeseen reasons or confounding reasons for DSRD symptoms at the study doctor's discretion.

Co-occurring Conditions

* Any co-occurring genetic disorder.
* Active symptomatic cardiac disease.
* Clinically significant chronic or active viral infection, including but not limited to HIV, hepatitis, CMV, EBV, HSV or untreated tuberculosis.
* Untreated chronic or active bacterial infection.
* Untreated hypothyroidism or hyperthyroidism.
* History of disseminated herpes zoster, disseminated herpes simplex, or recurrent localized dermatomal herpes zoster.
* History of malignancy (solid tumor or leukemia).
* Moyamoya syndrome or stroke (active or prior).
* Baseline abnormal renal function indicative of moderate or severe renal disease by eGFR <=45.
* History of acute narrow-angle glaucoma.
* History of venous or arterial thrombosis.
* IgA deficiency with antibodies against IgA.
* Pathogenic neuronal autoantibody positivity against established causes of autoimmune encephalopathy in CSF.
* Any subject with a history of anaphylaxis or a severe systemic response to blood or plasma-derived products.

Medications or Interventions

* Any vaccination planned during the study or within the last 6 weeks.
* Use of electroconvulsive therapy, lorazepam, or a JAK inhibitor within the last 4 weeks.
* Use of IVIG within the last 8 weeks.
* Use of immunosuppressant drugs (e.g., prednisone, mycophenolate mofetil, azathioprine) within the last 8 weeks.
* Use of rituximab within the past 6 months, unless B cell levels have recovered and are above 50 cells/uL.
* Use of other immunosuppressant biologics (e.g., adalimumab, etanercept) within the past 6 months.
* Use of strong CP3A4 inhibitors or inducers (e.g., ketoconazole, rifampin) within the last 4 weeks.
* Use of moderate CP3A4 inhibitors with a strong CYP2C19 inhibitor (e.g., fluconazole) within the last 4 weeks.
* Use of moderate CYP2C9 inhibitors (e.g., valproic acid) within the last 4 weeks.
* Use of strong CYP1A2 inducers (e.g., phenobarbital) or moderate CYP1A2 inhibitors (e.g., fluvoxamine) within the last 4 weeks.
* Use of certain mood stabilizers or anticonvulsants (e.g., clonazepam, lithium, oxcarbazepine) within the last 4 weeks.
* Any prior use of methotrexate, cyclophosphamide, or other chemotherapeutics.
* Any prior solid organ transplant.
* Any prior neurosurgical intervention.
* Any subject who has received blood or plasma products ≤ 30 days prior to first Baseline visit.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of number and severity of all adverse events. | Baseline to 14 weeks
  A summary of adverse events (AEs) by type and organ system will be reported for the entire study period, along with any statistically significant differences observed in rates of AEs across treatment arms.

SECONDARY OUTCOMES:
Change in catatonia by overall score in BFCRS. | Baseline to 12 weeks
  Change in overall score in the Bush-Francis Catatonia Rating Scale (BFCRS) between baseline and 12 weeks within or between treatment arms. A decrease in score indicates an improved performance.
Time to complete 25-Foot Walk assessment. | Baseline to 12 weeks
  Change in the time it takes to complete walking 25 feet between baseline to 12 weeks. A decrease in score indicates an improved performance.
Total number of errors in visual motor assessment NEPSY-II. | Baseline to 12 weeks
  Using NEPSY-II to measure change in total number of errors between both car and motorcycle trials. A decrease in score indicates an improved performance.
Change in expressive language as measured by total number of words used. | Baseline to 12 weeks
  Change in total number or words used in a guided language sample. An increase in score indicates improvement.
Change in adaptive skills as measured by the VABS-3 domain level standard score. | Baseline to 12 weeks
  Change in standard scores for at least one domain in the Vineland Adaptive Behavior Scales-3 (VABS-3) between baseline and 12 weeks within or between treatment arms. An increase in standard score by domain indicates improvement.
Change in family impact score as measured by summary score on PedsQL Family Impact Score. | Baseline to 12 weeks
  Change in the Pediatric Quality of Life Inventory (PedsQL) within or between treatment arms. An increase in summary score indicates improvement.
Change in quality of life score as measured by PedsQL summary score. | Baseline to 12 weeks
  Change in the Pediatric Quality of Life Inventory (PedsQL) summary score within or between treatment arms. An increase in summary score indicates improvement.

OTHER OUTCOMES:
Change in social interaction as measured by SRS-2 subdomain T-scores. | Baseline to 12 weeks
  Change in Social Responsiveness Scale-2 (SRS-2) subdomain treatment T-scores within or between treatment arms. A decrease in score indicates improvement.
Change in behavior as measured by DBC-2 T-score. | Baseline to 12 weeks
  A statistically significant change in Developmental Behavioral Checklist-2 (DBC-2) T-scores within or between treatment arms. A decrease in score indicates improvement.
Change in one or more measures of overall cognitive ability. | Baseline to 12 weeks
  A statistically significant change in one or more measures of overall cognitive ability within or between treatment arms.
  Measures include:
  * Behavior Rating Inventory of Executive Function, 2nd Edition (BRIEF-2): Change in T-scores.
  * Down Syndrome Mental Status Exam (DSMSE): Change in Total Memory and Non-Memory Composite score. .
  * Cambridge Neuropsychological Test Automated Battery (CANTAB) Paired Associate Learning (PAL) subdomain will be used to measure episodic learning.
  * CANTAB Spatial Span (SS) will be used to measure spatial processing.
  * CANTAB Reaction Time Interval (RTI) subdomain will be used to measure processing speed.
  * Kaufman Brief Intelligence Test-2 Revised (KBIT-2 Revised): Change in Standard Score.
  * Neuropsychiatric Inventory (NPI): Change in total score.
Change in receptive language as measured by PVT raw score. | Baseline to 12 weeks
  Change in the raw score of the NIH Toolbox Picture Vocabulary Test (PVT). An increase in score indicates an improved performance.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Espinosa, PhD, Principal Investigator — Linda Crnic Institute for Down Syndrome; Elise Sannar, MD, Principal Investigator — Children's Hospital Colorado; Jonathon Santoro, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be made available for all primary outcome measures.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available upon publication in a peer-reviewed journal.
Access Criteria: Data access requests will be reviewed by the sponsor-investigator and collaborators.